CLINICAL TRIAL: NCT04809961
Title: Longitudinal Observation of United Kingdom NHS Staff Wellbeing Following Introduction of the I-care Peer Support App
Brief Title: Longitudinal Observation of NHS Staff Wellbeing Following Introduction of the I-care Peer Support App
Acronym: I-Care
Status: Withdrawn | Type: Observational
Why Stopped: Recruitment
Sponsor: University of Southampton (Other)
Collaborators: Solent NHS Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 61764
Record Dates: First submitted 2021-02-02; First posted 2021-03-22 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Peer Group
Keywords: peer support; healthcare workforce; wellbeing; digital health; app
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: I-care app — A smart phone app to enable healthcare worker peer support for improved workplace wellbeing.

SUMMARY:
The coronavirus pandemic has had demonstrable impact upon healthcare workers. For healthcare workers this has meant disruption to vital access to peer support networks. In May 2020 the United Nations (UN) published a policy brief highlighting the importance of supporting mental health and wellbeing for communities affected by coronavirus. There is a need to find innovative solutions to facilitate support in the post-COVID-19 era and some innovations are emerging to fill this void but an evidence, long-term, sustainable, solution is yet to be proposed. In response, a digital app has been co-developed by UK researchers and healthcare staff with the intent to facilitate a virtual peer support mechanism for National Health Service (NHS) staff.

DETAILED DESCRIPTION:
Rationale: The coronavirus pandemic has had demonstrable impact upon healthcare workers. For healthcare workers this has meant disruption to vital access to peer support networks. In May 2020 the United Nations (UN) published a policy brief highlighting the importance of supporting mental health and wellbeing for communities affected by coronavirus. There is a need to find innovative solutions to facilitate support in the post-COVID-19 era and some innovations are emerging to fill this void but an evidence, long-term, sustainable, solution is yet to be proposed. In response, a digital app has been co-developed by UK researchers and healthcare staff with the intent to facilitate a virtual peer support mechanism for National Health Service (NHS) staff.

Aim: The main aim of this research is to determine the acceptability and efficacy of the newly developed I-care app to facilitate peer-support for NHS staff wellbeing.

Methods: A mixed methods study with concurrent process evaluation will be conducted to explore the acceptability and efficacy of an app-based peer support platform for use by anyone working within Solent NHS Trust with access to an android mobile phone device. Data will be generated from quantitative app usage, binary survey responses, and qualitative interviews.

Populations: All staff within Solent NHS Trust with an android mobile phone will be considered eligible to use the app.

Duration: Data will be collected at one, three, six, and 12-months post app launch.

Expected outcomes: As the innovation developed has spanned biomedical, behavioural and computing science a range of exploratory methods are proposed to establish the reach and uptake of the innovation, early indication of a potential causal model explaining how the innovation could lead to benefit, identification of key components of the innovation as identified by end users, and estimation of overall acceptability and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* All staff within a single UK Health Trust with an android mobile phone will be considered eligible to use the app

Exclusion Criteria:

* Not employed within the designated Trust
* Under 18 years of age
* Unable or unwilling to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All staff within a single UK Health Trust with an android mobile phone will be considered eligible to use the app.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Wellbeing | 12 months
  Most frequent response (A/B/C).

SECONDARY OUTCOMES:
Engagement | 12 months
  Number of participants who have provided a rating

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Cherry, PhD, Principal Investigator — University of Southampton & Solent NHS Trust
Locations (1):
- Lindsey Cherry, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No